CLINICAL TRIAL: NCT04005547
Title: Health Education and Relationships Through Theater: A Randomized Controlled Trial of Promoting Awareness Through Live Movement and Sound for Youth With Autism Spectrum Disorder (PALMS-ASD)
Brief Title: Health Education and Relationships Through Theater: An RCT of Promoting Awareness Through Live Movement and Sound for Youth With Autism Spectrum Disorder (PALMS-ASD)
Acronym: HEART
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: Public Health Management Corporation (Other)
Collaborators: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PublicHMC; 90AP2690-01-00 (Other Grant/Funding Number: Family and Youth Services Bureau)
Record Dates: First submitted 2018-04-13; First posted 2019-07-02 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Sexual Health; Education, Health
Keywords: sexual health; Autism Spectrum Disorders
MeSH Terms: conditions — Health Education; Autism Spectrum Disorder | interventions — Sound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program+survey (Experimental)
  Interventions: Behavioral: Promoting Awareness through Live Movement and Sound for youth with Autism Spectrum Disorder
- Survey-only (No Intervention)

INTERVENTIONS:
Behavioral: Promoting Awareness through Live Movement and Sound for youth with Autism Spectrum Disorder — Session 1 - Let's Talk About Relationships Session 2 - Let's Talk About Intimate Relationships Session 3 - Let's Talk About Sex Session 4 - Let's Talk About Protection Session 5 - Let's Talk About Communication *Bring your Trusted Adult* Session 6 - Let's Talk About Growing Up
  Other Names: PALMS-ASD
  Arms: Program+survey

SUMMARY:
Teens with ASD ages 14-19 will be screened for eligibility, complete a baseline interviewer/ACASI-administered survey, and randomly assigned to either intervention or control group. The enrollment goal is 500 teens. The 12-hour intervention will be run in groups of up to 12 teens, with health educators leading the group and actors assisting, role playing with participants, and performing a skit. Teens in the intervention group will take a post satisfaction survey, and teens in both conditions will take a 6-month and 12-month interviewer/ACASI-administered outcome survey. Fidelity will be monitored by observers and rated by health educators.

ELIGIBILITY:
Inclusion Criteria:

* meets age limits and
* parent/self-identifying as having an autism spectrum disorder, Asperger's Syndrome, or autism-similar social challenges, and/or
* mild intellectual disability

Exclusion Criteria:

* screen-out with screening tool, if not screened in by documented staff observation

  * Hospitalization within the last 3 months for a behavioral or mental cause
  * Inability to participate in group setting (sensory, extreme social/communication challenges)
  * Previous criminal conviction for sex offense
  * Sibling previously randomized to control
* screen-out with KBIT-2: Score < 50 OR Score above 70 on KBIT-2 and not receiving services for or having a diagnosis of ASD
* capacity to consent

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
unsafe sex self-report survey item | 6 months
  Frequency of condom with vaginal sex in past three months among those sexually active (none of the time, some of the time, all of the time). Will be reported if sufficient segment of sample is sexually active.
  PCM Q208. Have you EVER had vaginal sex? CMSEX
  PCM Q209. In the past three months, how many times did you have vaginal sex? CMVTIM
  Re-coded:
  PCM Q210. When you had vaginal sex in the past 3 months, how often did you or your partner use a condom? CMCNDM_R
  Response Options
  VSBO
  * CMSEX No, Yes, Refuse (0= No, 1=Yes, 8=RTA). CMVTIM 0 = I have never had sex
    1. = I have had sex but not in the past 3 months
    2. = Once in the past 3 months
    3. = 2-3 times in the past 3 months
    4. = 4 or more times in the past 3 months
    8 = Refuse to Answer
  * CMCNDM_R 1 'All of the time' .5 'Some of the time' 0 'None of the time' 8 'Missing'. (0= No, 1=Yes, 8=RTA).
unsafe sex self-report survey item | 12 months
  Frequency of condom with vaginal sex in past three months among those sexually active (none of the time, some of the time, all of the time). Will be reported if sufficient segment of sample is sexually active.
  PCM Q208. Have you EVER had vaginal sex? CMSEX
  PCM Q209. In the past three months, how many times did you have vaginal sex? CMVTIM
  Re-coded:
  PCM Q210. When you had vaginal sex in the past 3 months, how often did you or your partner use a condom? CMCNDM_R
  Response Options
  VSBO
  * CMSEX No, Yes, Refuse (0= No, 1=Yes, 8=RTA). CMVTIM 0 = I have never had sex
    1. = I have had sex but not in the past 3 months
    2. = Once in the past 3 months
    3. = 2-3 times in the past 3 months
    4. = 4 or more times in the past 3 months
    8 = Refuse to Answer
  * CMCNDM_R 1 'All of the time' .5 'Some of the time' 0 'None of the time' 8 'Missing'. (0= No, 1=Yes, 8=RTA).
sexual health knowledge self-report survey scale | 6 months
  sum of scored items (correct = 1/incorrect = 0): anatomy, STI prevention topics and pregnancy/birth control topics.
  Adapted from:
  National Survey of Reproductive and Contraceptive Knowledge Frost, Lindberg, & Finer, 2012 Healthy Oakland Teen Silver, & Bauman, 2006 National Survey of Adolescents and Young Adults National Longitudinal Adolescent to Adult Health Survey Rostosky, Regnerus, & Wright, "Coital Debut."
  Up to 33 questions scored, pending item psychometric performance (possible scale range 0 - 33)
adult-teen communication youth-report survey scale | 6 months
  comfort talking to a trusted adult about relationship/sexual health topics scale and/or having ever talked to a trusted adult about relationship/sexual health topics scale. Adapted for this study.
  Citation Sexual Health Communication Scale Jaccard, Dittus, & Gordon, 2000 Healthy Oakland Teen Silver, & Bauman, 2006 Scales TACT: Mean of 11 items based on talking to a trusted adult about (topic) and being told not to talk about something by a trusted adult (yes, no; none, some, all: mixed response options within scale - will be recoded, higher scores better) TACX/TACSE: mean of 5 items: i feel comfortable talking with a trusted adult (about topic), could you tell a trusted adult or talk with a trusted adult about (topic/event), 0- 19, 19 better
sexual health empowerment self-report survey scale | 6 months
  partner communication, boundary communication. Scale: Mean of 14 items. 0-19, score of 19 is better.
  Adapted for this study from Smylie et al., 2013; Silver, & Bauman, 2006
sexual health empowerment self-report survey scale | 12 months
  partner communication, boundary communication. Scale: Mean of 14 items. 0-19, score of 19 is better.
  Adapted for this study from Smylie et al., 2013; Silver, & Bauman, 2006
self-protective boundary knowledge self-report survey scale | 6 months
  knowledge of legality of sexual behaviors and knowledge of sexual/relationship behaviors reflecting being taken advantage of in a relationship. Created for this study. Scale: 7 items; Subscales: legal knowledge (5 items); power imbalance/being taken advantage of knowledge (2 items). All items scored as incorrect=0, correct=1. Scale score is average, which can be interpreted as percent correct.
self-protective boundary knowledge self-report survey scale | 12 months
  knowledge of legality of sexual behaviors and knowledge of sexual/relationship behaviors reflecting being taken advantage of in a relationship. Created for this study. Scale: 7 items; Subscales: legal knowledge (5 items); power imbalance/being taken advantage of knowledge (2 items). All items scored as incorrect=0, correct=1. Scale score is average, which can be interpreted as percent correct.

SECONDARY OUTCOMES:
sexual health efficacy self-report survey, item or scale | 6 months
  Sexual health self-efficacy Scale: Mean of 8 items. (condoms 3 items, birth control 2 items, STI testing 2 items, sexual health 1 item). 0-19, score of 19 is better.
  Condom scale (3 items) Acquiring condom self-efficacy 1 item (Q188) Adapted for this study from Smylie et al., 2013; Silver, & Bauman, 2006
sexual health efficacy self-report survey, item or scale | 12 months
  Sexual health self-efficacy Scale: Mean of 8 items. (condoms 3 items, birth control 2 items, STI testing 2 items, sexual health 1 item). 0-19, score of 19 is better.
  Condom scale (3 items) Acquiring condom self-efficacy 1 item (Q188) Adapted for this study from Smylie et al., 2013; Silver, & Bauman, 2006

OTHER OUTCOMES:
reasons for singleness | 6 months
  Strunz
  Q39. What prevents you from entering into a romantic relationship? Even if you are currently in a relationship, think about what prevented you from entering into a relationship before this.
  PREVREL What prevented a romantic relationship? 2 0 = Contact with others is too exhausting for me
  1. = I haven't yet met anybody with whom I could imagine having a romantic relationship
  2. = I am afraid of not fulfilling my partner's expectations
  3. = I don't know how to meet a potential partner
  4. = I don't know how a romantic relationship works or how to behave in a romantic relationship
  5. = I don't like the physical contact a romantic relationship brings with it
  6. = Sexual activities are unpleasant for me
  7. = I simply don't feel the need for a romantic relationship
  8. = Other reasons
  98 = Refuse to Answer
  Descriptives will be examined to create binary, categorical or dummy variables to examine impact on Response options 2 and 4.
reasons for singleness | 12 months
  Strunz
  Q39. What prevents you from entering into a romantic relationship? Even if you are currently in a relationship, think about what prevented you from entering into a relationship before this.
  PREVREL What prevented a romantic relationship? 2 0 = Contact with others is too exhausting for me
  1. = I haven't yet met anybody with whom I could imagine having a romantic relationship
  2. = I am afraid of not fulfilling my partner's expectations
  3. = I don't know how to meet a potential partner
  4. = I don't know how a romantic relationship works or how to behave in a romantic relationship
  5. = I don't like the physical contact a romantic relationship brings with it
  6. = Sexual activities are unpleasant for me
  7. = I simply don't feel the need for a romantic relationship
  8. = Other reasons
  98 = Refuse to Answer
  Descriptives will be examined to create binary, categorical or dummy variables to examine impact on Response options 2 and 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Management Corporation, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No